CLINICAL TRIAL: NCT05239702
Title: A Clinical Study on the Safety and Effectiveness of Targeting CD7 Chimeric Antigen Receptor T Cells in the Treatment of Autoimmune Diseases
Brief Title: Clinical Study of Targeting CD7 CAR-T Cells in the Treatment of Autoimmune Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, The President of The First Affiliated Hospital, College of Medicine, Zhejiang University, Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD7-002
Record Dates: First submitted 2021-12-01; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Crohn Disease; Ulcerative Colitis; Dermatomyositis; Still Disease; Autoimmune Diseases
Keywords: CAR T-cell therapy; CD7; Crohn disease; Ulcerative colitis; Dermatomyositis; Still disease; Refractory autoimmune disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Dermatomyositis; Arthritis, Juvenile; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Crohn Disease (Experimental)
  Interventions: Biological: CD7 CAR T-cells
- Ulcerative Colitis (Experimental)
  Interventions: Biological: CD7 CAR T-cells
- Dermatomyositis (Experimental)
  Interventions: Biological: CD7 CAR T-cells
- Still Disease (Experimental)
  Interventions: Biological: CD7 CAR T-cells
- Autoimmune Diseases (Experimental)
  Interventions: Biological: CD7 CAR T-cells

INTERVENTIONS:
Biological: CD7 CAR T-cells — Each subject receive CD7 CAR T-cells by intravenous infusion
  Other Names: CD7 CAR-T cells injection

SUMMARY:
A Clinical Study on the Safety and Effectiveness of Targeting CD7 Chimeric Antigen Receptor T Cells in the Treatment of Autoimmune Diseases

DETAILED DESCRIPTION:
Most patients with autoimmune diseases depend on hormones for life, and when poorly controlled, they are at risk of disability or even death. Studies have found that the abnormal T cell function of patients is closely related to the occurrence and development of the disease. Therefore, reducing the T cells in the patient's body or blocking the function has become the latest breakthrough in treatment. CD7 is a specific antigen on the surface of T cells. CD7 CAR-T can specifically attack T cells and has the potential to cure. In 2019, "Science Translational Medicine" magazine reported that the Marko Radic team demonstrated that CAR-T cells can achieve significant and long-lasting effects in the treatment of systemic lupus erythematosus (SLE) through animal experiments. In 2021, "NEJM" magazine reported the clinical efficacy of CAR-T cells in the treatment of SLE. In the same year, "Journal of Clinical Oncology" reported the clinical efficacy and safety of CD7 CAR-T cells in the treatment of T cell ALL.

Based on the current research status, we applied to clinical research on the treatment of refractory autoimmune diseases by targeting CD7 CAR-T cells. The selection criteria is patients with refractory autoimmune diseases. The purpose is to evaluate the safety and effectiveness of targeted CD7 CAR-T cell therapy through this clinical trial study, and to provide clinical evidence and experience reference for the application of CAR-T cell technology in the treatment of refractory autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as refractory Crohn disease, ulcerative colitis (collectively called Crohn's disease), and the conventional hormone therapy is not effective and (or) there is no effective treatment:

   1. At least 6 months before screening, diagnosed as Crohn's disease based on typical radiological results and/or typical histology.
   2. In addition to corticosteroids, after the use of immunosuppressive agents (usually azathioprine, methotrexate, and two biological agents (usually infliximab, adalimumab and/or setolizumab), the course of the disease is still Unsatisfactory. Patients should still have relapsed and refractory diseases after glucocorticoid and/or immunosuppressive treatment, or clearly show intolerance/toxicity to these drugs
2. Diagnosed as refractory dermatomyositis, and conventional hormone therapy is not effective and (or) ineffective treatment methods:

   1. At least 6 months before screening, confirmed or possible dermatomyositis according to Bohan and Peter criteria;
   2. At least it has no response to prednisone and other first-line immunosuppressants (such as methotrexate, mycophenolate mofetil, or azathioprine), or has obvious toxicity or intolerance to these therapies.
3. Refractory adult STILL disease

   1. Conform the diagnostic criteria for adult STILL disease (according to Yamaguchi et al., J. Rheumatology, 1992);
   2. After receiving non-steroidal anti-inflammatory drugs, glucocorticoids, anti-rheumatic drugs (DMARDs) and other treatments, there are still relapsed and refractory diseases, or clearly show that these drugs are intolerant/toxic.
4. Rheumatoid arthritis

   1. Conform the diagnostic criteria for rheumatoid arthritis in 2010 ACR classification criteria;
   2. Have received DMARDs or glucocorticoid therapy, but failed to achieve clinical remission, or clearly showed intolerance/toxicity to these drugs.

   The following screening can be performed by meeting any of the above 4 entry criteria
5. Estimated survival time> 12 weeks;
6. Patients had a negative urine pregnancy test before the start of administration and agreed to take effective contraceptive measures during the test period until the last follow-up;
7. Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

* Subjects with any of the following exclusion criteria were not eligible for this trial:

  1. History of craniocerebral trauma, conscious disturbance, epilepsy, cerebrovascular ischemia, and cerebrovascular, hemorrhagic diseases;
  2. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
  3. Pregnant (or lactating) women;
  4. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis);
  5. Active infection of hepatitis B virus or hepatitis C virus;
  6. Systemic steroids have used in the 4 weeks before participating in the treatment (except recently or currently using inhaled steroids);
  7. Those who have used any gene therapy products before.
  8. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
  9. Serum creatinine > 2.5mg/dl or ALT / AST > 3 times ULN or bilirubin > 2.0mg/dl;
  10. Those who suffer from other uncontrolled diseases are not suitable to join the study;
  11. HIV infection;
  12. Any situation that the researchers believe may increase the risk of patients or interfere with the test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Baseline up to 28 days after CD7 targeted CAR T-cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after CD7 targeted CAR T-cells infusion
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Overall response rate (ORR) | At Month 1, 3, 6, 12, 18, 24
  Proportion of subjects with complete or partial remission
Best overall response, BOR | At ≤3 month
  Assessment of ORR at ≤3 month
Concentration of CAR-T cells | From admission to the end of the follow-up, up to 2 years
  In peripheral blood and bone marrow
Duration of remission, DOR | 2 years post CD7 CAR-T cells infusion
  The time from the first assessment of remission or partial remission of the disease to the first assessment of disease progression or death from any cause
Overall survival (OS) | From CD7 CAR-T infusion to death，up to 2 years
  The time from the cell reinfusion to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China